CLINICAL TRIAL: NCT05075135
Title: Acceptability and Safety of 3D Printed Wrist-based Splints Compared to Plaster Casts for the Treatment of Non-surgical Distal Radius- and Scaphoid Fractures: a Randomized Feasibility Study.
Brief Title: Acceptability and Safety of 3D Printed Wrist-based Splints
Acronym: 3D-splinting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-00112
Record Dates: First submitted 2021-09-14; First posted 2021-10-12 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Distal Radius Fracture; Scaphoid Fracture
Keywords: 3D-splinting; Plaster cast; Patient satisfaction; Distal radius fracture; Scaphoid fracture
MeSH Terms: conditions — Wrist Fractures; Patient Satisfaction | interventions — Casts, Surgical

STUDY DESIGN:
Intervention Model Description: Randomization is based on a single allocation ratio of 1:1
  In order to generate an unpredictable allocation sequence and concealment of that sequence until assignment occurs, sequentially numbered, sealed, opaque envelopes will be prepared.
Masking Description: Masking is not feasible in this feasibility study, as the participants are not allowed to take off their splint (3D or plaster cast) during the bone healing time of 6 weeks. Care providers will take care of the patients prior to splint removal. Both the patients and the care providers are outcome assessors in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-splint group (Experimental): Patients wear the Swibrace 3D splint for 6 weeks of immobilization of the wrist for distal radius fractures, including the basis of the thumb for scaphoid fractures. X-rays after week 1, 3 and 6 are planned to document bone healing, together with weekly visits at the hand therapy unit to measure patient satisfaction and hand function. This results in 2-3 surgeon and 6 hand therapy visits at the Inselspital Bern, where regular check-ups on the patient's comfort in the splint are made.
  Interventions: Device: Swibrace 3D-splint
- Plaster cast group (Active Comparator): The control intervention is the same as the study intervention, but the participants wear the "gold-standard" plaster cast instead of the newly designed Swibrace 3D-splint.
  Interventions: Device: Plaster cast

INTERVENTIONS:
Device: Swibrace 3D-splint — The Swibrace 3D splint is a custom-made splint. For scanning of the forearms, the investigators will use the scanner "HandySCAN300" and the therewith delivered software "VXElements", the latter being necessary to create an accurate scan on the computer.
  Printing of the splint will be done by "Materialise", Belgium.
  Arms: 3D-splint group
Device: Plaster cast — The conservative gold standard treatment of distal radius and scaphoid fractures is applying a plaster cast. Therefore, patients in the control group follow standard therapy procedures.
  Arms: Plaster cast group

SUMMARY:
Non-invasiveness, avoidance of complications and comfort are important issues in the clinical management of conservatively treated distal radius and scaphoid fractures. To date, applying a plaster cast for approximately 6 weeks of immobilization is the gold standard. However, new 3D-technologies such as the design of Patient Specific Anatomical Braces (PSAB) will lead to a new paradigm of treatment. Swibrace has developed such anatomical, light, elegant and yet resistant braces. First, the fractured limb is scanned, the data then sent to a specifically designed software, printed in a 3D-printer and finally sent to the hospital for the patient's fitting. As these PSAB have not yet been tested on patients, the primary purpose of this study is to evaluate whether patient satisfaction with a 3D-printed PSAB differs from the one of traditionally treated patients in a plaster cast.

(A pre-clinical study will be conducted with 10 healthy volunteers testing the 3D splint for 72h. Only if splint satisfaction will be ≥ 70% as measured by the self-designed "Adult Rated Splint Evaluation Questionnaire" (ARSEQ), the 3D splint will be tested in patients. Otherwise, adjustments to the splint will be made based on the healthy volunteers' feedback prior to its testing in patients.)

DETAILED DESCRIPTION:
A criteria sample of 10 adult patients per group (Swibrace 3D splint and plaster cast) will be recruited in one University hospital in Switzerland and randomly assigned to either the 3D-splint or plaster cast group.

(For the pre-clinical study, the investigators aim to recruit 10 healthy volunteers testing one of the two 3D splint models (radius or scaphoid fracture splint).)

Study intervention:

Patients wear the Swibrace 3D splint for 6 weeks of immobilization of the wrist for distal radius fractures, including the basis of the thumb for scaphoid fractures. X-rays after week 1, 3 and 6 are planned to document bone healing, together with weekly visits at the hand therapy unit to measure patient satisfaction and hand function. This results in 2-3 surgeon and 6 hand therapy visits at the Inselspital Bern, where regular check-ups on the patient's comfort in the splint are made.

The control intervention is the same as the study intervention, but the participants wear the "gold-standard" plaster cast instead of the newly designed Swibrace 3D-splint. For the pre-clinical study, there is no control intervention.

(Healthy volunteers wear the Swibrace 3D splint for 72 hours. During this time, they are allowed to use their splinted hand for their usual daily activities, except for driving a car. They note their activities in a diary. At the end of the splint wearing time, they complete the ARSEQ. The scanning procedure will take at a place convenient for the volunteers.)

Study objectives:

The primary objective of this study is to assess if the patients' personal experiences and perceptions of safety and satisfaction (as defined by the self-designed "Patient rated splint evaluation questionnaire" (PRSEQ)) are superior in the Swibrace PSAB compared to a custom-made plaster cast.

Secondary objectives are:

To examine if there is a significant difference in self-perceived hand function and pain between the two groups (as assessed by the self-designed "Patient rated splint evaluation questionnaire" (PRSEQ)) To assess if radiological parameters between groups are similar at the end of the splint wearing period.

(To evaluate satisfaction with the 3D splint in healthy volunteers before testing the 3D splint in patients.)

The safety objectives are:

To document the attrition rate and - if applicable - reasons for drop-out in the Swibrace PSAB group (drop-out means that the participants make a cross-over to the control group until bone healing is assured) during the splint wearing time.

The X-ray appointments at Inselspital Bern, checking for the bone's correct healing position

The patients' safety perception (as assessed by the self-designed PRSEQ)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* ≥ 18 years old
* Understanding of German language (written and oral)
* Showing up at the Inselspital Bern emergency department with a stable, nondisplaced distal radius or scaphoid fracture that classifies a conservative immobilization treatment (as decided by the present surgeon on duty)

Exclusion Criteria:

* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* < 18 years old
* Vulnerable persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in "Patient Reported Splint Evaluation Questionnaire (PRSEQ)" | Part 1 will be filled out during (at week 2, 4, 6) and Part 2 after the splint wearing time (week 6).
  The investigators designed this questionnaire to the best of their knowledge due to lack of pre-existing orthosis satisfaction questionnaires suitable for the study purposes. The PRSEQ will be completed by the participating patients. It consists of two parts:
  Part 1 consist of 5 main topics: (1) pain because of the splint, (2) personal experiences with the splint, (3) personal safety, (4) specific and (5) usual activities in the splint. Pictures from the splint are given to allow ticking pressure marks and skin irritations where they appeared.
  Part 2 consists of 3 main topics: (6) satisfaction with the splint, (7) personal attitude and (8) satisfaction with the scanning procedure. Each main topic includes several sub-questions, where the patient rates his/her answers on a 11-point-Likert scale (0-10).

SECONDARY OUTCOMES:
Hand therapy evaluation - applying the "assessment of patient satisfaction" | Assessed during 6 hand therapy visits on a weekly basis until week 6, starting in week 1
  The assessment of patient satisfaction consists of 4 domains (patient comfort, patient compliance, cast odor and smell, skin itchiness) being rated on a 0-3 Likert Scale (0 = poor, 3 = excellent) by specialized hand therapists.
Hand therapy evaluation - finger range of motion as assessed by a hand-held goniometer | Assessed during 6 hand therapy visits on a weekly basis until week 6, starting in week 1
  The hand-held goniometer will be used to measure the distances between the finger tips and the palm of the hand in centimeters. A touch-down (finger tips touch the palm) will be judged with "yes/no". Both finger range of motion measurements will be assessed by specialized hand therapists.
Hand therapy evaluation - sensibility as measured by the "Ten Test" | Assessed during 6 hand therapy visits on a weekly basis until week 6, starting in week 1
  Specialized hand therapists will assess sensibility by applying the quantitative sensory test "Ten Test". The patient reports his/her light touch perception of the skin area being tested compared to the reference normal area when the examiner (hand therapist) gives a simultaneous stimulus by stroking a normal area and the area under examination. The response from the patient rating the sensibility of the test area is recorded as a fraction out of 10 between 1/10 and 10/10 (10 = normal sensory perception).
Hand therapy evaluation - pain as measured by the "Numeric Rating Scale" | Assessed during 6 hand therapy visits on a weekly basis until week 6, starting in week 1
  Specialized hand therapists will assess pain using the Numeric Rating Scale for pain. It requires the patient to rate their pain on a defined scale from 0-10, where 0 is no pain and 10 is the worst pain imaginable. Patients are asked to circle their current pain in their hand on this scale.
Bone position - x-ray evaluation by specialized hand surgeons and orthopedists | 2-3 regular x-rays will take place during the bone healing phase after 1 week of splint wearing, if necessary in week 2 and after 6 weeks as assessed by physicians
  Bone healing process is closely monitored by specialized hand surgeons and orthopedists by taking an x-ray on several time points:
  - one week after the accident to check if the bone is not displaced to guarantee that a conservative treatment may be continued.
  in case of any uncertainties, another x-ray will take place during week 2 after the accident to check on the bone's position again.
  - after 6 weeks, the last x-ray will be made to decide removal of the plaster cast / 3D splint
Questionnaire "assessment of clinical effectiveness" as rated by specialized hand surgeons and orthopedists | Administered once at the end of the study after 6 weeks
  The "assessment of clinical effectiveness" is an assessment where 4 domains are judged by specialized hand surgeons or orthopedists on a 0-3 Likert Scale (0 = poor, 3 = excellent). These are: stability of immobilization, blood circulation, wear pressure-related pain and pressure sores.
Composite endpoint "adherence" assessed as the "number of clinical visits that were missed" / "number of drop-outs" and "number of patients crossing over to the plaster cast group" | Ongoing during the whole study period of 6 weeks
  Adherence will be documented by clinicians (hand therapists and physicians) in terms of counts of: clinical visits that have taken place (or being missed), drop-out or cross-over rates to the plaster cast group.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Vögelin, Prof, Study Director — Department of Plastic and Hand Surgery (DOPH)
Locations (1):
- Inselspital Bern, Hand therapy research unit, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study description at Inselspital Bern, Switzerland — http://servicenow.insel.ch/studien?id=ins_studien_form&table=u_contract_management&sys_id=e8ae7960ec6d741046e96abb57855137
- See also: collaboration partner, 3D-technology, Fribourg, Switzerland — http://www.swibrace.com/
- See also: 3D printing company, Belgium — https://www.materialise.com/en/about